CLINICAL TRIAL: NCT01490853
Title: Long Term Follow-up of Ph+ CML Patients Achieving Complete Cytogenetic Remission With Interferon Based Therapy
Brief Title: Follow-up of Ph+ Chronic Myleoid Leukemia Patients in Complete Cytogenetic Response With Interferon Based Therapy
Status: Completed | Type: Observational
Sponsor: Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Domenico Russo, Director, Università degli Studi di Brescia
Other Study IDs: CML0509
Record Dates: First submitted 2011-12-01; First posted 2011-12-13 (Estimated); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Ph pos CML; Philadelphia positive Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- CML and interpheron alpha: Adult Ph+CML pts in CCgR after IFN alpha.
  Interventions: Drug: Interpheron alpha

INTERVENTIONS:
Drug: Interpheron alpha — Long term outcom after interferon alpha discontinuation or not

SUMMARY:
Objectives

This is an observational study aimed at updating the overall survival (OS), the progression free survival (PFS) to accelerated-blastic (AB) phase and the complete cytogenetic response (CCgR) duration of the CML patients who between 1986 and 2001 were treated with an IFN based therapy (either alone or in combination) and who obtained a CCgR. It also aims at analysing the clinical and biological features of this selected cohort of patients with persisting CCgR after treatment with IFN.

Study design This study is an observational retrospective multicenter study.

Assessment and Follow-up Patients' demographic data and retrospective collection of CML cytogenetic and molecular data will be reported in the "Assessment and Follow-up FORM".

In this FORM the events related to therapy, disease and survival will also be reported.

Duration of the study:

The recruitment period is estimated in approximately 2 years.

DETAILED DESCRIPTION:
Study rational

* IFN, either alone or in combination with AC, prolonged survival of Ph+ CML patients, in early chronic phase, mainly in those patients achieving the CCgR
* CCgR became the surrogate marker for survival duration and the main target of IFN therapy
* CCgR were rare events accounting for less than 10% of the cytogenetic responsive patients
* These cases can be considered as a fascinating elite of patients who have the highest sensitivity to IFN and are the most likely candidates for prolonged survival and possibly cure
* From 1986 to 2001, more than 1200 CML patients either enrolled in different national trials or referred in single Institutions have been treated frontline with IFN based therapy
* In 2001, data on 317 CCgRs were reported by the EICML group
* They included 214 cases treated with IFN alone collected from the database of 9 national study groups in Austria, Belgium, Netherlands, France, Germany, Italy, Spain, Sweden and United Kingdom and 103 cases treated with IFN alone collected from single Institutions in Italy, France, and United Kingdom.
* The study did not include the patients achieving CCgR with IFN + LDAC
* The contribution of Italy was of 119 cases: 59 from national studies and 60 from single Institutions
* The follow-up of these patients is stopped at 2000 and from 2000 thereafter almost CML patients were treated with IM
* We don't know if the patients who had achieved a CCgR with IFN based therapy continued or discontinued IFN, or crossed to IM therapy
* We don't know if they maintained a CCgR with or without therapy
* We don't know if the patients who achieved a CCgR with IFN and crossed to IM had the same cytogenetic and molecular response, PFS and OS as the majority of the patients unresponsive to IFN who were treated with IM
* We don't know the clinical and biological features of these selected cohort of patients

ELIGIBILITY:
Inclusion criteria

* Age > 18 years
* Ph+/BCR-ABL+ CML in CP
* Treatment with IFN alpha alone or in combination ( i.e HU, Ara-C, YNK01, ASCT ), either within or outside national Study Protocols.
* Complete cytogenetic response (CCgR) (0% Ph+ cells)
* Written informed consent prior to any study procedures being performed.

Exclusion Criteria:

* Patients with Ph+ CML in accelerated/blastic phase (AP/BP)
* No treatment with Interferon-alpha
* No written informed consent prior to any study procedures being performed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (>18 years old) patients with CP Ph+/BCR-ABL CML and with CCgR after therapy including IFN alpha.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2009-10; Primary Completion 2012-01 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | From date of enrollment until the date of first documented progression, assessed up to 240 months
  One primary outcome measure is the PFS of the CML patients who between 1986 and 2001 were treated with IFN based therapy (either alone or in combination) and who obtained the CCgR.
Duration of Complete Cytogenetic Response (CCgR) | From date of enrollment until the date of first documented loss of CCgR, assessed up to 240 months
  One primary outcome measure is the duration of CCgR of the CML patients who between 1986 and 2001 were treated with IFN based therapy (either alone or in combination) and who obtained the CCgR.
Overall Survival | From date of enrollment until the date of first documented death from any cause, assessed up to 240 months
  OS will be calculated from the date of diagnosis until date of death (whatever the cause). Patients still alive will be censored at the moment of last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Domenico Russo, Study Director — Università degli Studi di Brescia
Locations (1):
- Chair of hematology, Brescia, Italy